CLINICAL TRIAL: NCT02433886
Title: Efficacy and Adverse Events of Bilateral Single-shot Ventral Capsular/Ventral Striatal Gamma Capsulotomy for Obsessive-compulsive Disorder: a Pilot Study
Brief Title: Efficacy and Adverse Events of Bilateral Single-shot VC/VS Gamma Capsulotomy for OCD: a Pilot Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Hospital do Coracao (Other); Brown University (Other)
Responsible Party: Principal Investigator, Antonio Carlos Lopes, Antonio Carlos Lopes MD, PhD, University of Sao Paulo General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GammaOCD_IPq_HCor
Record Dates: First submitted 2015-04-29; First posted 2015-05-05 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-04

CONDITIONS: Obsessive-compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gamma Ventral Capsulotomy (Experimental)
  Interventions: Procedure: Gamma Ventral Capsulotomy

INTERVENTIONS:
Procedure: Gamma Ventral Capsulotomy
  Other Names: Ventral capsular/ventral striatal gamma capsulotomy

SUMMARY:
Up to 40% of Obsessive-Compulsive Disorder (OCD) patients do not respond to conventional treatments (medications or behavior therapy). For some of them, a neurosurgical treatment can be indicated. A previous study, employing bilateral double-shot ventral capsular/ventral striatal (VC/VS) Gamma capsulotomy (GVC) for OCD has shown that this radiosurgical technique is potentially efficacious and relatively safe. However, a few patients may develop complications associated to radionecrosis (eg., brain cysts) in a long-term follow-up, which are probably associated to lesion volumes. Another study, with the preliminary results of smaller VC/VS Gamma capsulotomy lesions has suggested that this procedure is safe and remains efficacious. Our aim is to investigate the efficacy and safety profiles of smaller, single-shot VC/VS Gamma capsulotomy for OCD. This study will support the development of a future double-blind, randomized clinical trial of single-shot VC/VS Gamma capsulotomy.

ELIGIBILITY:
Inclusion Criteria:

* A DSM-V diagnosis of OCD as the main diagnostic entity. If comorbid axis I or II disorders are present, OCD symptoms are the most troublesome among disorders.
* Age range between 18 and 65 years old.
* At least 5 years of OCD symptoms.
* "Yale-Brown Obsessive-Compulsive Scale" (YBOCS) scores greater than 26 (or greater than 13, for isolated obsessions or compulsions).
* Refractoriness criteria fulfilled.
* To be accepted by the "best estimate" method as a treatment refractory patient. It consists in the careful examination of each patient's history by two OCD specialists, so as to confirm refractoriness status.

Refractoriness criteria:

* At least 3 serotonin reuptake inhibitors (selective or not) have been tried before. One of these trials must have included clomipramine. All drugs were used for a minimum of 12 weeks, at the maximum doses or the maximally tolerated doses.
* Previous participation in a cognitive behavior therapy program (exposure and response prevention), for a minimum of 20 hours' time; or participation for some time, without subsequent adherence, due to severe OCD symptoms, and acceptance of the independent review board.
* YBOCS scores reductions after adequate drug therapy and psychotherapy not better than 25 %, or confirmation of no clinical improvements by the mental health professionals who were responsible for the treatments of the patient.
* By the end of adequately conducted pharmacological trials, "Clinical Global Impression" (CGI) scores not better than minimal improvement.
* Previous use of at least two antidepressant augmentation strategies (such as the association of a typical or atypical antipsychotic, another serotonin reuptake inhibitor, a benzodiazepine, an anticonvulsant or an antiglutamatergic medication), in adequate doses for a sufficient period of time, without satisfactory responses.

Exclusion Criteria:

* Less than 18 years or more than 65 years of age.
* Past history of head injury, with posttraumatic amnesia.
* Past or general medical condition, or neurological illness with brain compromise (severe and in active phase)
* History of physiological effects of a substance, as determinant of psychopathological symptoms, or cumulative signs of alcohol or drug abuse in the Central Nervous System (such cortical atrophy), confirmed by a neuroimaging scan.
* Pregnancy or lactation.
* Refusal to participate in radiosurgical procedures.
* Refusal to sign the Patient Information and Consent Form, or refusal to take part in this study.
* History of mental retardation and/or being unable to understand the Patient Information and Consent Form, confirmed by poor performance on neuropsychological tests.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2014-12; Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | up to 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- OCD Clinics (PROTOC), Department of Psychiatry, University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil